CLINICAL TRIAL: NCT01817153
Title: Effect of Intravenous Hydrocortison on Post-ischemic Brachial Artery Dilation and on Thenar Oxygen Saturation in Adult Septic Shock. A Human Placebo-controlled Randomized Study.
Brief Title: Effect of Hydrocortison on Post-ischemic Flow-mediated Dilation and on Thenar Oxygen Saturation in Human Septic Shock.
Acronym: HyStOON
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: not enough recruitment
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Principal Investigator, Thierry BOULAIN, M.D., Centre Hospitalier Régional d'Orléans
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHRO-2012-04; 2012-004736-39 (EudraCT Number)
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Septic Shock; Adult
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): 10 mL normal saline iv at H0 and H6 (2 first injections blinded), followed by hydrocortison (open label) 50 mg iv at H8, H14 and H20
  Interventions: Drug: placebo followed by hydrocortisone hemisuccinate
- hydrocortison (Active Comparator): 50 mg hydrocortison iv at H0 and H6 (2 first injections blinded), followed by hydrocortison (open label) 50 mg iv at H12, H18 and H24
  Interventions: Drug: hydrocortison hemisuccinate

INTERVENTIONS:
Drug: hydrocortison hemisuccinate
  Arms: hydrocortison
Drug: placebo followed by hydrocortisone hemisuccinate
  Arms: placebo

SUMMARY:
The main objectives of the study are 1)to examine the immediate (2 hours) and delayed (8 hours) effects of intravenous hydrocortison on macro and microvascular post-ischemic vasoreactivity, in septic shock adult patients; 2) to examine possible correlations between post-ischemic flow-mediated dilation (FMD) of the brachial artery (assessed by ultrasound imaging) and post-ischemic recovery slope of the thenar oxygen saturation (StO2) (assessed by near-infrared spectroscopy).

DETAILED DESCRIPTION:
Two primary end points, considered as reflecting vasoreactivity will be assessed :

1. Flow-mediated dilation (FMD) of the brachial artery, measured by ultrasound imaging, expressed in mm or in percentage, will be calculated from artery diameters measured before and after a vascular occlusion test (cuff around arm or forearm).
2. recovery slope of thenar oxygen saturation (StO2), assessed by near infrared spectroscopy (NIRS), expressed in %/second, will be recorded after the vascular occlusion test.

The two primary end points (FMD and recovery slope of StO2)will be assessed at the following timepoints :

* baseline (before first injection of placebo or hydrocortison)
* 2 hours after first injection of placebo or hydrocortison
* 2 hours after second injection of placebo or hydrocortison (i.e. 8 hours after first injection)
* 4 to 6 hours after third injection
* 4 to 6 hours after fourth injection (optional)

ELIGIBILITY:
Inclusion Criteria:

* age over 18 yrs
* consent obtained
* septic shock (according to international definition)
* patient sedated and submitted to invasive mechanical ventilation
* no need for surgery expected within 24 hours after enrollment
* patient has received at least one dose of large spectrum antibiotics
* superior vena cava catheter in place
* patient carrying a thermodilution device for cardiac output measurement
* stable mean arterial pressure within 65-5 mmHg limits for at least 2 hours;

Exclusion Criteria:

* pregnancy
* age below 18 years
* patient treated with iv continuous epinephrine
* chronic occlusive arteriopathy of the upper limbs
* regular or recent treatment with glibenclamide or glipizide
* regular or recent treatment with steroids
* known surrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Vasoreactivity | every 6 hours over the first 24 hours of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Boulain, MD, Principal Investigator — Centre Hospitalier Régional d'Orléans, France
Locations (1):
- Centre Hospitalier Régional d'Orléans, Orléans, France